CLINICAL TRIAL: NCT07388082
Title: Total Laparoscopic vs Open Pancreaticoduodenectomy for the Treatment of Periampullary Adenocarcinomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mahmoud Rady, Lecturer of general surgery, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT (670)
Record Dates: First submitted 2025-12-07; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Periampullary Carcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional open pancreaticoduedectomy (Active Comparator): 15 patients underwent conventional open pancreaticoduedenctomy
  Interventions: Procedure: Conventional open pancreaticoduedectomy
- Total laparoscopic pancreaticoduedectomy (Active Comparator): 15 patients underwent total laparoscopic pancreaticoduedectomy
  Interventions: Procedure: Total laparoscopic pancreaticoduedectomy

INTERVENTIONS:
Procedure: Conventional open pancreaticoduedectomy — Fifteen patients in Group A had a traditional open pancreaticoduedectomy.
  Arms: conventional open pancreaticoduedectomy
Procedure: Total laparoscopic pancreaticoduedectomy — Fifteen patients in Group A had a total laparoscopic pancreaticoduedectomy.
  Arms: Total laparoscopic pancreaticoduedectomy

SUMMARY:
Laparoscopic pancreaticoduodenectomy (LPD), a surgical option for nonpancreatic periampullary adenocarcinoma (NPPA), is a complex procedure that has become increasing popular. However, there is no consensus as to whether this technique should be performed routinely. Our aim was to evaluate the outcomes of LPD compared with open pancreaticoduodenectomy (OPD).

ELIGIBILITY:
Inclusion Criteria:

* • Body mass index <28.0 kg/m2.

  * Ampullary tumors, duodenal tumors restricted to the second part of the duodenum, or lower common bile duct tumors.
  * Carefully confirmed resectability of the tumors based on preoperative radiology conducted by experienced radiologists and surgeons.

Exclusion Criteria:

* • Patients with >180 degrees superior mesenteric artery encasement

  * Any celiac abutment.
  * Unreconstructable superior mesenteric vein/portal occlusion" Aortic invasion or encasement.
  * A history of previous upper abdominal surgery.
  * Tumors extending to the uncinate.
  * Severe cardiorespiratory comorbidities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-05 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-10-05 (Actual)

PRIMARY OUTCOMES:
The incidence of pancreatic fistula after laparoscopic pancreaticoduodenectomy in comparison to open surgery | in 2 years between 2023 - 2025
  Laparoscopic pancreaticoduodenectomy is a complex procedure that has become increasing popular. However, there is no consensus as to whether this technique should be performed routinely.
  Our aim was to evaluate the outcomes of Laparoscopic pancreaticoduodenectomy compared with open pancreaticoduodenectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paniccia A, Schulick RD, Edil BH. Total Laparoscopic Pancreaticoduodenectomy: A Single-Institutional Experience. Ann Surg Oncol. 2015 Dec;22(13):4380-1. doi: 10.1245/s10434-015-4450-2. Epub 2015 Apr 18. PMID 25893407